CLINICAL TRIAL: NCT04651010
Title: Predictive Multimodal MRI Factors in Subacute Cerebral Artery Occlusiontreated by Thrombectomy (PIMISUTT
Brief Title: Predictive Multimodal MRI Factors in Subacute Cerebral Artery Occlusiontreated by Thrombectomy (PIMISUTT)
Acronym: PIMISUTT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Poitiers University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: PIMISUTT; 2020-A021118-31 (Registry Identifier: ID-RBC)
Record Dates: First submitted 2020-11-25; First posted 2020-12-03 (Actual); Last update posted 2024-12-16 (Actual); Status verified 2024-12

CONDITIONS: Middle Cerebral Artery Acute Ischemic Stroke
Keywords: Ischemic stroke; acute middle cerebral artery occlusion; multimodal MRI; thrombectomy
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Multimodal MRI (Experimental)
  Interventions: Other: Multimodal MRI

INTERVENTIONS:
Other: Multimodal MRI — Multimodal MRI will be realized between 12 and 24 hours after thrombectomy

SUMMARY:
Our study aims to measure metabolic and functional parameters of the infarcted territory by multimodal cerebral MRI in patients diagnosed with unilateral proximal occlusion of the middle cerebral artery and treated by thrombectomy in order to correlate those parameters to clinical outcome (evaluated by modified Rankin score) at 3 months.

We aim to find early radiologic predictive factors for favorable clinical outcome in this population of patients.

DETAILED DESCRIPTION:
The treatment of acute ischemic stroke in the setting of intracranial large artery occlusion and especially middle cerebral artery occlusion (MCAO) with intravenous tissue plasminogen activator (IV-tPA) is associated with low rates of recanalization and high rates of neurological morbidity and functional dependence.

In the last few years, endovascular intervention (mechanical thrombectomy) has proven its safety and its efficacy on clinical outcome in patients diagnosed with MCAO and is now commonly recommended.

However, in this population of patients treated by thrombectomy, very few predictive factors, except for the post-procedural recanalization score (TICI), do exist to foresee the variability of clinical outcome.

Tissue viability of the infarcted territory can be approached by the measure of metabolic and morphological parameters (Na+, H+, phosphore, diffusion imaging) which can be non-invasively done by multimodal MRI, as suggest by recently published studies.

Our study plans to measure these parameters between 12 and 24 hours after acute ischemic stroke in patients with MCAO treated by thrombectomy in order to correlate those parameters to clinical outcome at 3 months (modifier Rankin Score).

ELIGIBILITY:
Inclusion Criteria:

* Patients aged ≥ 18 years old
* Hospitalized at the Poitiers University Hospital
* Acute middle cerebral artery occlusion diagnosed by CT-scan or MRI
* NIHSS score ≥ 6 at admission
* To be treated by thrombectomy with or without fibrinolysis
* Written information delivered to the patient or his relatives concerning the study and its benefit and risk

Exclusion Criteria:

* Patients or relatives whom a loyal information about the study cannot be given
* Patient with cognitive impairments before MRI.
* Patients who cannot undergo MRI because of contraindications
* Patients too deteriorated to tolerate one hour long exam

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2021-11-15 (Actual); Primary Completion 2025-08-15 (Estimated); Study Completion 2025-08-15 (Estimated)

PRIMARY OUTCOMES:
Correlation between modified Rankin score at 3 months and multimodal MRI data | Month 3

SECONDARY OUTCOMES:
Discharge National Institute of Health Stroke Score (NIHSS) | Month 3
National Institute of Health Stroke (NIHSS) score at 3 months | Month 3
Change in NIHSS score at 3 months compared to post-thrombectomy | Month 3

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Poitiers, Poitiers, France

IPD SHARING:
Plan to Share IPD: Undecided